CLINICAL TRIAL: NCT04119362
Title: PARAGON Platform for Outcome, Quality of Life, and Translational Research on Pancreatic Cancer
Acronym: PARAGON
Status: Completed | Type: Observational
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: PARAGON; AIO-LQ-0214 (Other: Arbeitsgemeinschaft Internistische Onkologie)
Record Dates: First submitted 2019-09-25; First posted 2019-10-08 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: pancreas; quality of life; PRO; Pancreatic Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples With DNA — Formalin Fixed and Paraffin Embedded Tumor Tissue (FFPE)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pancreatic adenocarcinoma: Patients with metastatic pancreatic cancer receiving will be asked to fill in an EORTC QLQ-C30 questionnaire and additional questionnaires on worries about quality of life impairments and physical constitiution every 8 weeks, over the entire course of treatment, starting with neo-/adjuvant or 1st line therapy follow. There is no restriction on type of therapy. No further intervention.
  Interventions: Other: Quality of live questionnaires; Other: Optional translational project

INTERVENTIONS:
Other: Quality of live questionnaires — EORTC-Q30 questionnaire, additonal questionnaire on worries about quality of life impairments and on physical condition every 8 weeks. No additional visits will be carried out for questionnaires. Questionnaires will be handed out to patients during routine visits.
Other: Optional translational project — Collection of archival tumor material for future translational projects. No biopsy will be performed in the context of this registry. Only tumor samples obtained in the context of standard of care and after explicit informed context will be used.

SUMMARY:
Due to the generally poor prognosis, with no chance of long-term survival, health related quality of life is a very important objective in the treatment of patients with pancreatic cancer. The non-interventional, prospective, multicentre PARAGON study is desinged to evaluate the health-related quality of life in patients with metastatic pancreatic cancer, by analyzing the course of QoL throughout all applied therapy lines for patients with pancreatic adenocarcinoma, measured according to EORTC scoring manual and patient reported outcome.

DETAILED DESCRIPTION:
Pancreatic cancer is often diagnosed at an advanced stage, because most of the patients have no symptoms until the cancer metastasized. In the majority of study cases pancreatic cancer research focuses on therapy outcomes and prognosis. With poor prognosis and no chance of long-term survival, quality of life becomes a very significant purpose of pancreatic cancer care.

The PARAGON study is designed to see a bigger picture by acquiring data on quality of life (QoL) and further outcome of patients with localized, locally advanced and metastatic pancreatic cancer and moreover to establish a sample collection for future biomarker analysis.

The multicenter, prospective, permanent, register study PARAGON collects outcome data, patient reported outcomes (PRO), and tumor tissues of pancreatic cancer patients of both sexes and ages over 18 at approx. 80 German study sites. Patients diagnosed with pancreatic adenocarcinoma planned for (or recently started with) neoadjuvant, adjuvant or 1st line therapy can be included into the study.

The data assessment includes data on demography, basic parameters, anamnesis, comorbidities, therapies, outcome and survival data as well as patient reported outcome in QoL at baseline and every 8 weeks.

PARAGON's first objective is to determine the course of QoL throughout all applied therapy lines for patients with pancreatic adenocarcinoma, measured according to EORTC scoring manual and patient reported outcome. Secondary outcome measurements are e.g. progression-free, disease-free and overall survival according to treatment line.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and signed data protection form before any study specific intervention, including screening, will be done
* Age ≥ 18 years
* Histologically or cytologically confirmed pancreatic adenocarcinoma
* Systemic neoadjuvant, adjuvant, 1st line systemic therapy is planned or recently started (within last 14 days)

Exclusion Criteria:

* Patients who are unable to consent because they do not understand the nature, significance and implications of the study
* Patients who are unable to understand or fill out the QoL survey
* Patients in 2nd or further treatment lines that have not been documented for 1st line therapy within the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The course of Quality of Life (QoL) throughout the entire course of therapy for patients with pancreatic adenocarcinoma | through study completion, an average of 1 year
  EORTC-QLQC30 according to EORTC scoring manual
Other patient reported outcome (PRO) | through study completion, an average of 1 year
  Physical performance status patient questionnaire according to ECOG criteria

SECONDARY OUTCOMES:
Progression- free survival (PFS) | through study completion, an average of 1 year
  As for the main objective, there is no formal secondary endpoint in a registry study. Therfore, in this section we will explain the main data to be collected and the main outcome measures.
Disease-free survival (DFS) | through study completion, an average of 1 year
  As for the main objective, there is no formal secondary endpoint in a registry study. Therfore, in this section we will explain the main data to be collected and the main outcome measures.
Overall survival (OS) | through study completion, an average of 1 year
  As for the main objective, there is no formal secondary endpoint in a registry study. Therfore, in this section we will explain the main data to be collected and the main outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof., Study Director — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest; Thorsten Goetze, Prof., Principal Investigator — Krankenhaus Nordwest gGmbH Institut für Klinisch-Onkologische Forschung; Ralf Hofheinz, Prof., Principal Investigator — Universitätsmedizin Mannheim
Locations (24):
- Germany (24):
  - HELIOS Klinikum Bad Saarow, Bad Saarow
  - MVZ am Oskar-Helene-Heim, Berlin
  - Klinikum Coburg, Coburg
  - Onkozentrum Dresden/Freiberg, Dresden
  - Gemeinschaftspraxis Hämatologie und Onkologie, Erfurt
  - Institute for Clinical Cancer Research Krankenhaus Nordwest, Frankfurt
  - Klinikum Frankfurt Höchst, Frankfurt
  - Universitätsklinikum Halle, Halle
  - Überörtliche Gemeinschaftspraxis Schwerpunkt Haematologie, internistische Onkologie & Palliativmedizin, Hamburg
  - St. Bernward Krankenhaus, Hildesheim
  - Klinikum Kassel Klinik für Hämatologie und Onkologie, Kassel
  - Klinikum Konstanz, Konstanz
  - ÜBAG - MVZ Dr. Vehling-Kaiser GmbH Hämatologisch-onkologische Tagesklinik Landshut, Landshut
  - Magdeburg, Klinikum Magdeburg gGmbH, Magdeburg
  - Mayen, Institut für Versorgungsforschung, Mayen
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Hämatologisch-Onkologische Schwerpunktpraxis, Naunhof
  - Friedrich-Ebert-Krankenhaus, Neumünster
  - medius KLINIK OSTFILDERN RUIT, Ostfildern
  - BAG Innere Medizin - Hämatologie - Onkologie, Regensburg
  - Elblandklinikum Riesa, Riesa
  - RoMed Klinikum Onkologische Tagesklinik, Rosenheim
  - Onkologische Schwerpunktpraxis, Speyer
  - Marienhospital, Stuttgart

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.